CLINICAL TRIAL: NCT07188987
Title: Bilateral Sphenopalatine Ganglion Block Using Prilocaine Versus Lidocaine as Adjuvants to General Anesthesia During Endoscopic Hypophysectomy, Randomized Trial.
Brief Title: Prilocaine for Sphenopalatine Ganglion Block in Endoscopic Hypophysectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Rania Samir Fahmy, Associate professor, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MS- 403-2021
Record Dates: First submitted 2025-08-28; First posted 2025-09-23 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-09

CONDITIONS: Blood Pressure Control
Keywords: Sphenopalatine ganglion block; Prilocaine; lidocaine; endoscopic hypophysectomy
MeSH Terms: interventions — Lidocaine; Sphenopalatine Ganglion Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Lidocaine (L) (Active Comparator): Group L will receive 2ml of 2% lidocaine and 0.5ml of diluted adrenaline.
  Interventions: Procedure: Sphenopalatine Ganglion Block using 2% lidocaine
- Group Prilocaine (P) (Experimental): Group P will receive 2ml of 4% prilocaine and 0.5ml saline
  Interventions: Procedure: Sphenopalatine Ganglion Block
- Group Prilocaine adrenaline (PA) (Experimental): Group PA will receive 2ml of 4% prilocaine and 0.5ml of diluted adrenaline.
  Interventions: Procedure: Sphenopalatine Ganglion Block

INTERVENTIONS:
Procedure: Sphenopalatine Ganglion Block using 2% lidocaine — Sphenopalatine ganlion block with 2ml of 2% lidocaine and 0.5ml of diluted adrenaline after general anesthesia in patients undergoing enoscopic hypophysectomy.
  Arms: Group Lidocaine (L)
Procedure: Sphenopalatine Ganglion Block — Sphenopalatine ganlion block with will receive 2ml of 4% prilocaine and 0.5ml saline after general anesthesia in patients undergoing enoscopic hypophysectomy.
  Arms: Group Prilocaine (P)
Procedure: Sphenopalatine Ganglion Block — Sphenopalatine ganlion block with will receive 2ml of 4% prilocaine in addition to 0.5ml of diluted adrenaline. after general anesthesia in patients undergoing enoscopic hypophysectomy.
  Arms: Group Prilocaine adrenaline (PA)

SUMMARY:
Patients undergoing endoscopic surgeries for pituitary adenoma excision suffer from wide swings in blood pressure that might increase bleeding and interfere with the surgical field.

Local anethetic infiltration and regional nerve blocks have been used to provide better analgesia, control blood pressure and improve surgical field.

Limited studies evaluated shenopalatine ganglion block in pituitary adenoma excision with promising outcomes. The proposed study will compare the efficacy of two local anesthetics, prilocaine and lidocaine, for spenopalatine ganglion block in patients undergoing endoscopic pituitary adenoma excision. Evaluating the control of the intraoperative blood pressure and analgesic sparing are the main objectives of the proposed study.

DETAILED DESCRIPTION:
Pituitary adenoma excision through endoscopic sinus surgery has been evolving over the years. Though less traumatic less traumatic and less invasive than other approaches, hemodynamic variations during several phases of the surgey as nasal dissection pose challenges for anesthesiologists.

Regional techniques present appealing options for better control of blood pressure during periods of maximal surgical stimulation, they may as well provide a better surgical field. One of the regional techniques is the sphenopalatine ganglion bock where a local anesthetic is injected in the pterygopalatine fossa around the sphenopalatine ganglion. Thus, It blocks pain transmission through the branches of the trigeminal nerve.

The current study was designed to compare the effects of two local anesthetics, lidocaine versus prilocaine on intraoperative hemodynamics, surgical field and analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pituitary adenoma undergoing endoscopic hypophysectomy.
* ASA physical status I and II.
* Age above 21, below 45 years.
* Male or female

Exclusion Criteria:

* Any patient below 21 years or above 45 years.
* Patients suffering from any of the following conditions:

  * Disturbed conscious level.
  * Coagulation abnormalities.
  * Poorly controlled blood pressure and/or heart rate.
  * Increased intracranial tension.
  * Liver and kidney disorders.
* Patients on anticoagulants and/or NSAIDS (non-steroidal anti- inflammatory drugs
* Patients addicted to drugs and/or alcohol.
* Patients with disturbed conscious level at the end of the surgery, GCS >14

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
MAP | Mean arterial blood pressure in mmhg in the intraoperative period 5 minutes after nasal dissection
  mean arterial blood pressure in the intraoperative period 5 minutes after nasal dissection
MAP | Mean arterial blood pressure in mmhg after 5 minutes of nasal dissection
  mean arterial blood presssure 5 minutes after nasal dissection

SECONDARY OUTCOMES:
Mean arterial blood pressure | Before induction of Anesthesia, Before the block, 15 minutes after the block, 5 min of nasal dissection and every 30 minutes till the end of operation.
  Mean arterial blood pressure in mmhg before induction of Anesthesia, Before the block, 15 minutes after the block, 5 min of nasal dissection and every 30 minutes till the end of operation.
Systolic blood pressure | Systolic blood pressure in mmhg before induction of Anesthesia, Before the block, 15 minutes after the block, 5 min of nasal dissection and every 30 minutes till the end of operation.
  Systolic blood pressure before induction of Anesthesia, Before the block, 15 minutes after the block, 5 min of nasal dissection and every 30 minutes till the end of operation.
Diastolic blood preesure | Diastolic blood pressure in mmhg before induction of Anesthesia, Before the block, 15 minutes after the block, 5 min of nasal dissection and every 30 minutes till the end of operation.
  Diastolic blood pressure before induction of Anesthesia, Before the block, 15 minutes after the block, 5 min of nasal dissection and every 30 minutes till the end of operation.
HR | Heart rate in beats/min before induction of Anesthesia, Before the block, 15 minutes after the block, 5 min of nasal dissection and every 30 minutes till the end of operation.
  Heart rate before induction of Anesthesia, Before the block, 15 minutes after the block, 5 min of nasal dissection and every 30 minutes till the end of operation.
Patients needing propranolol | The number of patients throughout the study in the intraoperative period who received propranolol
  The number of patients needing propranolol in each group.
Propranolol needed | The amount of propranolol in mg used throughout the surgery in each group
  The total amount of propranolol in mg used in each group
Patients needing phentolamine | The number of patients receiving phentolamine throughout the surgery in both groups
  The number of patients needing phentolamine in each group.
Phentolamine needed | Throughout the surgical time from the begining to the end of surgery
  The total amount of phentolamine in mg used in each group.
Surgeon satisfaction scale | 10 minutes after the end of surgery.
  Surgeon satisfaction scale based on Average category scale (ACS) from 0 to 5 with 0 meaning no bleeding and 5 massive uncontrollable bleeding
Time to 1st analgesic requirement | The time in hours from emergence of anaesthesia till the request of first rescue analgesia in the first 24 hours after surgery
  The time from emergence of anaesthesia till the request of first rescue analgesia
Blood loss | Throughout the surgical time from the begining to the end of surgery
  The total ammount of blood loss in cc
Requirement for transfusion | Throughout the surgical time from the begining to the end of surgery
  The number of patients requiring transfusion
Fentanyl needed | Throughout the surgical time from the begining to the end of surgery
  number of patients needing fentanyl boluses intraoperatively
Total amount of fentanyl | Throughout the surgical time from the begining to the end of surgery
  total ammount of fentanyl needed in micrograms

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The detailed protocol describing the techniques used in the study and the anesthetic conduct and the outcome measures.
  The statistical plan to analyze the different outcome measures.
Supporting Information: Study Protocol, SAP
Time Frame: IPD can be available 3 months after completion of the study
Access Criteria: IPD can be accessed from the authors by journals considering the study for publication and upon reasonable request from other investigators

REFERENCES:
- [Background] Chaudhary R, Payal YS, Mohapatra B, Sony S, Shekhar S. USG-guided bilateral sphenopalatine ganglion block: A useful anesthetic adjuvant for trans nasal trans sphenoidal pituitary surgery in a patient with severely low ejection fraction. Saudi J Anaesth. 2025 Jan-Mar;19(1):102-104. doi: 10.4103/sja.sja_388_24. Epub 2025 Jan 1. PMID 39958315
- [Background] Rezaeian A, Hashemi SM, Dokhanchi ZS. Effect of Sphenopalatine Ganglion Block With Bupivacaine on Postoperative Pain in Patients Undergoing Endoscopic Sinus Surgery. Allergy Rhinol (Providence). 2019 Jan 23;10:2152656718821282. doi: 10.1177/2152656718821282. eCollection 2019 Jan-Dec. PMID 30719401
- [Background] Cafiero T, Cavallo LM, Frangiosa A, Burrelli R, Gargiulo G, Cappabianca P, de Divitiis E. Clinical comparison of remifentanil-sevoflurane vs. remifentanil-propofol for endoscopic endonasal transphenoidal surgery. Eur J Anaesthesiol. 2007 May;24(5):441-6. doi: 10.1017/S0265021506002080. Epub 2007 Mar 12. PMID 17376252
- [Background] Jane JA Jr, Thapar K, Kaptain GJ, Maartens N, Laws ER Jr. Pituitary surgery: transsphenoidal approach. Neurosurgery. 2002 Aug;51(2):435-42; discussion 442-4. PMID 12182782